CLINICAL TRIAL: NCT01332617
Title: Phase II Study of Simvastatin, Zoledronic Acid, Bortezomib, Bendamustine and Methylprednisolone for Relapsed/Refractory Myeloma
Brief Title: Phase II Study of Simvastatin for Relapsed/Refractory Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators no longer interested in activating study
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-HEM-10-001
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Simvastatin; Zoledronic; Bortezomib; Bendamustine; Methylprednisolone
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Simvastatin; Methylprednisolone; Bortezomib; Diclofenac; Bendamustine Hydrochloride; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with combination therapy (Experimental): Treatment with combination therapy of Simvastatin, Zoledronic Acid, Bortezomib, Bendamustine, and Methylprednisolone.
  Interventions: Drug: Simvastatin,Zoledronic Acid,Bortezomib,Bendamustine,Methylprednisolone.

INTERVENTIONS:
Drug: Simvastatin,Zoledronic Acid,Bortezomib,Bendamustine,Methylprednisolone. — 1. Simvastatin 80 mg PO daily starting day -2 through day 10.
  2. Zoledronic acid 4 mg IV over 15 minutes on day 1 and then monthly
  3. Bortezomib 1.3 mg/m2/day IV bolus on days 3,6 and 10.
  4. Bendamustine 100 mg/m2/day IV over 30 minute infusion on days 3 and 10.
  5. Methylprednisolone 1g/m2 IV over 30 minutes on days 1 and 8.
  Other Names: Simvastatin (ZOCOR); Methylprednisolone (Medrol); Bortezomib (Voltarol, Diclofenac); Bendamustine (Treanda); Zoledronic acid (Zometa, Reclast, Zomera)

SUMMARY:
The purpose of this study test the hypothesis that the combination of simvastatin and zoledronic acid (for reversal of drug resistance), with bortezomib, high-dose methylprednisolone and bendamustine on a day 1,8 schedule (to reduce toxicity) will be an effective and well-tolerated treatment for relapsed and refractory multiple myeloma

DETAILED DESCRIPTION:
OBJECTIVES

Primary To estimate the overall response rate (ORR) (complete response (CR) + very good partial response (VGPR) + partial response (PR)) of patients with multiple myeloma who have relapsed or are refractory after bortezomib treatment and will now receive a combination therapy of simvastatin, zoledronic acid, bortezomib, bendamustine and methylprednisolone.

To evaluate safety and tolerability of studied therapy.

Secondary

1. To estimate the progression-free Survival (PFS), time to progression (TTP), overall survival (OS) and duration of response (DOR).
2. To describe toxicities (frequency and severity) during the treatment. 3 To estimate clinical benefit response (CBR) (ORR + minor response (MR)) and stable disease (SD).

4 Explore factors associated with ORR, PFS, OS, toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Multiple Myeloma (using the International Myeloma Working Group Guidelines)
* Patients must have failed at least one prior treatment regimen containing bortezomib.

They may be refractory to primary therapy or relapsed and have measurable or assessable disease. (Refractory disease is defined as anything less than PR or progression within 60 days of completing therapy.)

* Patients with Multiple Myeloma must have measurable active, progressive or symptomatic disease. Measurable disease may be paraprotein or free light chains in serum or urine, or the presence of bone marrow plasma cells.
* Age- must be at least 18 years of age.
* Prior therapies may include bendamustine, bortezomib, methylprednisolone, radiation, and autologous hematopoietic cell transplant.
* Patients who have received therapy must be at least 4 weeks beyond prior chemotherapy (excluding corticosteroids).
* If female patient with reproductive capacity: on effective means of birth control during the entire duration of the treatment.
* Patients must have recovered from acute toxicities resulting from therapy administered prior to entering this study to grade 1 or less. Alopecia may not be resolved.
* Ability to understand and willingness to sign a written informed consent document.
* Life expectancy of greater than 8 weeks.
* ECOG performance status 0, 1, or 2 (Karnofsky > 60%; see Appendix A).
* Patients must have adequate bone marrow function as defined below:

absolute neutrophil count > 500/ul platelets > 30,000/ul

-Patients must have adequate liver function as defined below: total bilirubin < 2 times the upper limit of normal AST(SGOT), ALT(SGPT) < 3 x upper limit of normal

* Patients must have adequate renal function as defined by a creatinine clearance > 40 mL/min (measured or estimated by the Cockcroft-Gault formula).
* Patients must have no signs of significant rhabdomyolysis determined by CPK levels with a CK < 5 times the upper limit of normal.

Exclusion Criteria:

* Patients who have not received any chemotherapy treatment for multiple myeloma prior to being enrolled in the study.
* Patients who were receiving simvastatin (dose > 40 mg/day), or the equivalent dose of another statin) during last prior chemotherapy for multiple myeloma.
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients receiving any other investigational agent(s).
* Active second malignancy in the last 5 years except for non-melanoma skin cancer or carcinoma-in-situ.
* History of hypersensitivity reactions attributed to simvastatin, bortezomib, bendamustine or zoledronic acid.
* Pregnant women are ineligible, as treatment involves unforeseeable risks to the embryo or fetus.
* Patients receiving medications that may increase risk of rhabdomyolysis such as itraconazole, ketoconazole, erythromycin, cyclosporine, amiodarone, verapamil, niacin, HIV protease inhibitors.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myopathy, untreated hypothyroidism, hereditary myopathy in the family history, unstable angina pectoris, liver disease not due to multiple myeloma, cardiac arrhythmia that is symptomatic or not rate controlled, active connective tissue disease, active autoimmune disease, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Response to treatment as defined by The International Myeloma Working Group response criteria for multiple myeloma. | 4 weeks after first dose of simvastatin
  Response catergories (IMWG):
  Complete Remission(CR), Very Good Partial Remission(VGPR), Partial Remission (PR), Minor Response (MR), Progressive Disease (PD), Stable Disease, Relapse,Refractory Disease, Overall Response.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | After 1 year of follow-up.
  PFS is measured from date of study enrollment until the date of progressive disease is documented.
Incidence Rate of Toxicity | End of study; monitoring during study.
  Decriptive statistics will be provided regarding incidence rates of toxcity. Patients will be monitored for safety throughout the study.
Overall Survival (OS) | After 1 year of follow-up
  OS is measured from date of study enrollment until death.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Herzig, MD, Principal Investigator — James Graham Brown Cancer Center- University of Louisville